CLINICAL TRIAL: NCT00851149
Title: Pro-inflammatory Cytokines (IL-1beta,IL-6, IL-8 and TNF-α) and Complement Activation (C3a) in Blood Collected From Surgery Field From Patients Undergoing Orthopedic Surgery Compared to Patients Undergoing Abdominal Aneurysm Repair.
Brief Title: Pro-inflammatory Cytokines in Blood From Orthopedic Surgery Compared to Abdominal Aneurysm Repair
Acronym: KEEP-HB
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sykehuset i Vestfold HF (Other)
Collaborators: Oslo University Hospital (Other); Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Espen Lindholm/Consultant, Hospital in Vestfold HF
Other Study IDs: 6.2009.36
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Aortic Diseases; Osteoarthritis, Hip
Keywords: aorta; disease; abdominal; surgery; Osteoarthritis, Hip; replacement; blood; autolog; transfusion; cytokines
MeSH Terms: conditions — Aortic Diseases; Osteoarthritis, Hip; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1/10: Abdominal aortic surgery patients
  Interventions: Device: Sangvia blood sampling system
- 2/10: Total hip replacement patients
  Interventions: Device: Sangvia blood sampling system

INTERVENTIONS:
Device: Sangvia blood sampling system — Blood collected from abdominal aortic repair patients are compared against blood collected from total hip replacement patients
  Other Names: Sangvia Blood Salvage System

SUMMARY:
The purpose of this study is to investigate the contents in blood sampled from surgery site during hip replacement compared with blood sampled from abdominal aortic surgery. Is there any difference in pro-inflammatory cytokines (IL-1beta, IL-6, IL-8 and TNF-α), complement activation (C3a)?

DETAILED DESCRIPTION:
Patient (n= 10) scheduled for total hip replacement or hemiprosthesis and patient (n=10) scheduled for abdominal aortic surgery.

Primary outcome:

Pro-inflammatory cytokines (IL-6, IL-8 and TNF-α) and complement activation (C3a) in blood samples collected from surgery field. Comparison between the 2 groups.

Secondary outcome:

Haemoglobin, Trc, INR in blood samples and plasma will be analysed and compared between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-4

Exclusion Criteria:

* Patient using corticosteroids, NSAIDs or Cox-II inhibitors
* Patients under 18 years
* Patients who are included in pharmaceutical studies
* Opioids-, benzodiazepines-, antiepileptic drugs-, alcohol- and α2-agonists abuse
* Pregnant and breastfeeding women
* Patients with known hypersensitivity for opioids, propofol or volatile anesthetics
* Patients with serious arrhythmias (atrial fibrillation/flutter is acceptable)
* Uncontrolled hypertension, serious psychiatric disease
* Patients with unstable angina pectoris or myocardial infarction the last month before inclusion
* Acute abdominal aortic surgery (acute dissection or rupture)
* Planned laparoscopic abdominal aortic aneurysm surgery
* Transfusion of blood products last month before surgery
* Glucocorticoid users

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-02 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Pro-inflammatory cytokines (IL-6, IL-8 and TNF-α) and complement activation (C3a) in blood samples collected from surgery field. Comparison between the 2 groups. | 30 days

SECONDARY OUTCOMES:
Haemoglobin, Trc, INR in blood samples and plasma will be analysed and compared between the 2 groups. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Espen Lindholm, Md, Principal Investigator — Sykehuset i Vestfold HF
Locations (1):
- Sykehuset i Vestfold HF, Tønsberg, Norway